CLINICAL TRIAL: NCT03282071
Title: Community-based Mental Wellness Project for Adolescents and Adults: Joyful Parenting Pilot Project RCT Study
Brief Title: Joyful Parenting Pilot Project RCT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Family Welfare Society (Other)
Responsible Party: Principal Investigator, Dr Sun Yuying, Post-doctoral Fellow, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPH-MHP-FWS01
Record Dates: First submitted 2017-09-06; First posted 2017-09-13 (Actual); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Mental Well-being; Happiness
Keywords: Mental health; Mental well-being; Community-based engagement; Positive psychology; Public health approach
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Joyful Parenting Intervention (Experimental): Subjects will participate in two-session interactive talks on joyful parenting (a core session intervention and booster intervention) and one family gathering activity; questionnaire evaluation will be conducted at baseline, post-session,1 month and 3 month after core session.
  Interventions: Behavioral: Joyful Parenting Intervention
- Control (No Intervention): No intervention will be provided to control groups during study period.

INTERVENTIONS:
Behavioral: Joyful Parenting Intervention — * Two-session interactive talks for parents to promote praise & appreciation, positive thinking, enjoyable parenting (mind) and knowledge of adult mental health problem (in particular the mixed anxiety and depressive disorder) and mental well-being.
  * One family gathering activity (e.g. outdoor / visit / family indoor gathering) to promote and practise quality family communication (enjoyment and sharing).
  Arms: Joyful Parenting Intervention

SUMMARY:
Aims: To enhance mental well-being of adolescents, adults and their families by creating a positive, happy and joyful environment in the community.

Targets: Parents aged 12-59 and their family members in Hong Kong.

Methods: Joyful Parenting Pilot Project will adopt the public health and family-focused approach, under the brand name of "Joyful@HK Campaign". Evidence-based and Evidence Generating approach with vigorous study design, both qualitative (e.g. focus groups) and quantitative (e.g. randomised controlled trial), will be used to evaluate the overall programme effectiveness including follow-up of at least one month ("best science"). To ensure the practicability and sustainability of the CBEP, we will engage community partners with strong track records of "best practice" to design, plan, and implement the intervention. This project will use innovative and integrated positive psychology and public health theories and methods to plan brief, simple, and cost-effective intervention.

Significance: By using "best science" in the design and evaluation of intervention programme, and the "best practice" of the partners' skills, experience and strong connection with service targets in the community, the intervention, if proven to be effective, for promoting sharing, mind and enjoyment and enhancing mental wellbeing can be further developed and widely disseminated to and adopted by the practitioners in the health and social service sectors for replication and improvement to benefit the whole population.

DETAILED DESCRIPTION:
Joyful Parenting Pilot Project is part of the Community-based Mental Wellness Project for Adolescents and Adults, which aims at enhancing mental well-being of adolescents, adults and their families by creating a positive, happy and joyful environment in the community. The Project is funded by Health Care and Promotion Fund of Food and Health Bureau.

Joyful Parenting Pilot Project is organized by the Hong Kong Family Welfare Society and led by the School of Public Health, The University of Hong Kong (HKU). The project will organize two-session interactive talks for parents to promote praise and appreciation, positive thinking, enjoyable parenting and knowledge of adult mental health problem (in particular the mixed anxiety and depressive disorder) and mental well-being; and one family gathering activity to promote and practice quality family communication. One wisdom sharing session will be organized for social workers and service practitioners to promote best practice of community mental wellness project.

The major subjects of the Joyful Parenting Pilot Project RCT Study are 120 parents and at least 240 family members. 4 family service units of Hong Kong Family Welfare Society will either be assigned into intervention groups or wait-list control groups. Cluster Randomized Controlled Trial will be used to evaluate the effectiveness of the intervention programme.

In the study, parents and their family members will be invited to complete questionnaires to measure the behavioral indicators of sharing, mind and enjoyment, and mental well-being and/or invited to attend the focus group to understand the participants' experience during the programme while community partners will be invited to individual in-depth interviews. HKU team will conduct evaluation during the programme implementation stage. The effectiveness of the intervention, as well as the level of participation and ratings for the intervention will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Parents (major subjects):

   * Parents aged 18-59 (including single parents)
   * Chinese speaking
   * Able to complete questionnaires/ focus groups
2. Their family members:

   * Family members of those parents who have already participated in the Joyful Parenting Pilot Project (Their family members could be children/ adolescents)
   * Chinese speaking
   * Able to complete questionnaires/ focus groups
3. Community partners

   * Staff of Integrated Family Service Units, under Hong Kong Family Welfare Society in partnership with HKU research team, who organize, plan or implement the project
   * Adults aged 18 or above
   * Chinese speaking
   * Able to complete questionnaires/ individual in-depth interviews

Exclusion Criteria:

* Those who cannot read Chinese
* Those who suffered from severe mental illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuying Sun, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Hong Kong Family Welfare Society- North Point Integrated Family Service Centre, Hong Kong
  - Hong Kong Family Welfare Society- Yau Tong Integrated Family Service Centre, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun Y, Wang MP, Chan CS, Lo DLO, Wan ANT, Lam TH, Ho SY. Promoting positive parenting and mental wellbeing in Hong Kong Chinese parents: A pilot cluster randomised controlled trial. PLoS One. 2022 Jul 20;17(7):e0270064. doi: 10.1371/journal.pone.0270064. eCollection 2022. PMID 35857769

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: Aug-Oct 2017; types of location: family service centres
Pre-assignment Details: 8 parents excluded (not meeting inclusion criteria 18-59 years)
Units Other Than Participants: family service centres
Groups:
- Joyful Parenting Intervention: Two sessions of interactive talks were included with each lasted for 2 hours. The contents included praise and appreciation skills, enjoyable parenting through family games and knowledge of Mixed Anxiety and Depressive Disorder (MADD).
  After around 3 months, a family gathering activity also involving the children and other family members was organized as an incentive for the parents.
- Control: No intervention were provided to control groups during assessment period.
Period: Overall Study
Arm/Group | Joyful Parenting Intervention | Control
Started | 75; 2 family service centres | 69; 2 family service centres
Completed | 65; 2 family service centres | 60; 2 family service centres
Not Completed | 10; 0 family service centres | 9; 0 family service centres

BASELINE CHARACTERISTICS:
Groups:
- Control: No intervention were provided to control groups during study period.
- Total: Total of all reporting groups
Arm/Group | Joyful Parenting Intervention | Control | Total
Number analyzed (Participants) | 75 | 69 | 144
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 41.8 (5.51) | 43.3 (6.19) | 42.5 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 64 | 122
  Male | 17 | 5 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Birthplace [Number; unit: participants]
  Hong Kong | 28 | 27 | 55
  Guangdong Province | 29 | 27 | 56
  Other places | 18 | 15 | 33

OUTCOME MEASURES:

1. Primary Outcome: Sharing (Praise), Mind (Appreciation) and Enjoyment (SME) Related Behaviours
Description: Outcome-based questionnaire will be used to evaluate participants' frequency of performing the suggested Sharing, Mind and Enjoyment (SME) related behaviours from baseline to three-month after baseline.
  Praise: 3-item (range: 0-21). Higher scores mean a better outcome. Appreciation: 2-item (range: 0-14). Higher scores mean a better outcome. Enjoyment: 2-item (range: 0-14). Higher scores mean a better outcome.
Time Frame: T1: baseline; T3: 1-month follow-up after baseline; T4: 3-month follow-up after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Joyful Parenting Intervention | Control
Number analyzed (Participants) | 75 | 69
score on a scale
  Sharing (Praise) at baseline | 11.49 (5.15) | 11.34 (4.79)
  Sharing (Praise) at 1-month | 12.23 (4.91) | 11.05 (4.81)
  Sharing (Praise) at 3-month | 13.09 (4.12) | 12.34 (4.22)
  Mind (Appreciation) at baseline | 7.03 (3.72) | 7.86 (3.56)
  Mind (Appreciation) at 1-month | 8.37 (3.66) | 8.44 (3.36)
  Mind (Appreciation) at 3-month | 8.86 (2.81) | 7.83 (2.91)
  Enjoyment at baseline | 7.78 (3.78) | 7.42 (3.29)
  Enjoyment at 1-month | 7.82 (3.22) | 7.58 (3.09)
  Enjoyment at 3-month | 8.92 (3.31) | 7.75 (2.77)

2. Secondary Outcome: Changes in Subjective Happiness From Baseline to Three-month After Baseline
Description: Subjective Happiness Scale (4 items) (1-7): higher scores mean a better outcome.
Time Frame: T1: baseline; T3: 1-month follow-up after baseline; T4: 3-month follow up after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: No intervention will be provided to control groups during assessment period.
Arm/Group | Joyful Parenting Intervention | Control
Number analyzed (Participants) | 75 | 69
score on a scale
  Subjective Happiness at baseline | 4.47 (1.19) | 4.52 (1.10)
  Subjective Happiness at 1-month | 5.03 (1.10) | 4.54 (1.08)
  Subjective Happiness at 3-month | 5.12 (0.93) | 4.64 (1.05)

3. Secondary Outcome: Changes in Mental Well-being From Baseline to Three-month After Baseline
Description: Validated Chinese version of 7-item Warwick Edinburgh Well-being Scale (7-35): higher scores indicated higher level of wellbeing.
Time Frame: T1: baseline; T3: 1-month follow-up after baseline; T4: 3-month follow up after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Joyful Parenting Intervention | Control
Number analyzed (Participants) | 75 | 69
score on a scale
  Mental well-being at baseline | 24.82 (3.8) | 23.82 (4.62)
  Mental well-being at 1-month | 25.81 (3.94) | 24.67 (3.74)
  Mental well-being at 3-month | 27.32 (3.83) | 24.81 (4.55)

4. Secondary Outcome: Changes in Family Relationship From Baseline to Three-month After Baseline
Description: Respondents rated each item from 0 (no understanding / intimacy / communication at all with family members) to 10 (full understanding / intimacy / communication with family members), resulting in a total score of 0-30, with higher scores indicating better family relationship.
Time Frame: T1: baseline; T3: 1-month follow-up after baseline; T4: 3-month follow up after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Joyful Parenting Intervention | Control
Number analyzed (Participants) | 75 | 69
score on a scale
  Family relationship at baseline | 20.71 (6.80) | 20.85 (5.05)
  Family relationship at 1-month | 22.36 (5.03) | 20.73 (4.76)
  Family relationship at 3-month | 23.06 (4.69) | 20.34 (5.23)

5. Secondary Outcome: Changes in Personal and Family Health From Baseline to Three-month After Baseline
Description: Respondents rated each item from 0 (not at all healthy) to 10 (very healthy), with higher scores indicating higher level of personal/family health.
Time Frame: T1: baseline; T3: 1-month follow-up after baseline; T4: 3-month follow up after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Joyful Parenting Intervention | Control
Number analyzed (Participants) | 75 | 69
score on a scale
  Personal health at baseline | 6.15 (2.05) | 6.10 (2.27)
  Personal health at 1-month | 6.99 (2.04) | 6.18 (2.23)
  Personal health at 3-month | 7.29 (1.84) | 6.32 (2.15)
  Family health at baseline | 6.25 (2.32) | 6.25 (2.22)
  Family health at 1-month | 7.23 (1.87) | 6.48 (1.94)
  Family health at 3-month | 7.33 (1.66) | 6.50 (1.95)

6. Secondary Outcome: Changes in Personal and Family Happiness From Baseline to Three-month After Baseline
Description: Respondents rated each item from 0 (not at all happy) to 10 (very happy), with higher scores indicating higher level of personal/family happiness.
Time Frame: T1: baseline; T3: 1-month follow-up after baseline; T4: 3-month follow up after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Joyful Parenting Intervention | Control
Number analyzed (Participants) | 75 | 69
score on a scale
  Personal happiness at baseline | 6.15 (2.31) | 6.15 (2.19)
  Personal happiness at 1-month | 6.97 (1.99) | 6.45 (2.11)
  Personal happiness at 3-month | 7.25 (1.79) | 6.37 (2.07)
  Family happiness at baseline | 6.40 (2.54) | 6.37 (2.13)
  Family happiness at 1-month | 7.38 (1.99) | 6.55 (1.92)
  Family happiness at 3-month | 7.45 (1.67) | 6.46 (1.98)

7. Secondary Outcome: Changes in Family Harmony From Baseline to Three-month After Baseline
Description: Respondents rated each item from 0 (not at all harmonious) to 10 (very harmonious), with higher scores indicating higher level of family harmony.
Time Frame: T1: baseline; T3: 1-month follow-up after baseline; T4: 3-month follow up after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Joyful Parenting Intervention | Control
Number analyzed (Participants) | 75 | 69
score on a scale
  Family harmony at baseline | 6.23 (2.59) | 6.49 (2.09)
  Family harmony at 1-month | 7.20 (2.09) | 6.80 (1.96)
  Family harmony at 3-month | 7.39 (1.89) | 6.63 (1.96)

8. Secondary Outcome: Changes in Knowledge and Perception of Mixed Anxiety and Depressive Disorders
Description: The knowledge and understandings of MADD was self-developed to assess the level of awareness of the MADD symptoms ("I know the symptoms of MADD", range 0 to 10), intention to seek help ("I will talk to families or friends when I have emotional disturbance", range 0-10), self-efficacy of help seeking ("I know how to seek help when I have emotional disturbance", range 0-10), and understanding of the MADD definition ("MADD refers to the condition when both anxiety and depression are diagnosed", yes/no/uncertain).
Time Frame: T1: baseline; T3: 1-month follow-up after baseline; T4: 3-month follow up after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Joyful Parenting Intervention | Control
Number analyzed (Participants) | 75 | 69
score on a scale
  The awareness of MADD symptoms at baseline | 4.85 (2.61) | 5.30 (2.74)
  The awareness of MADD symptoms at 1-month | 7.33 (1.81) | 4.95 (2.90)
  The awareness of MADD symptoms at 3-month | 7.23 (2.07) | 5.50 (2.61)
  Intention to seek help at baseline | 6.28 (2.44) | 7.05 (2.49)
  Intention to seek help at 1-month | 7.47 (1.88) | 7.18 (2.21)
  Intention to seek help at 3-month | 7.72 (1.95) | 7.14 (2.25)
  Self-efficacy at baseline | 6.94 (2.36) | 7.07 (2.47)
  Self-efficacy at 1-month | 7.50 (2.01) | 7.24 (2.16)
  Self-efficacy at 3-month | 7.89 (1.99) | 7.04 (2.35)

9. Secondary Outcome: Satisfaction Towards Joyful Parenting Intervention Programme
Description: Satisfaction towards programme will be assessed by program evaluation measures: rated on a 0-10 scale, with "0" indicating "unsatisfied" and "10" indicating "satisfied".
Time Frame: T2: after 1st talk; T3: 1-month follow-up after baseline; T4: 3-month follow up after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Joyful Parenting Intervention
Number analyzed (Participants) | 75
score on a scale
  Satisfaction of the 1st talk at T2 | 8.47 (1.44)
  Satisfaction of the 2nd talk at 1-month | 8.48 (1.29)
  Satisfaction of the family gathering at 3-month | 8.80 (1.17)

ADVERSE EVENTS:
Time Frame: No adverse event was observed at post-intervention (T2), 1-month (T3) or 3-month (T4).
Arm/Group | Joyful Parenting Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/69
Other Adverse Events (participants affected / at risk) | 0/75 | 0/69

LIMITATIONS AND CAVEATS:
Validated questionnaires were not available and many existing questionnaires were too long, we developed the outcome and impact-oriented questionnaires to assess the changes in the participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT03282071/Prot_SAP_000.pdf